CLINICAL TRIAL: NCT06807034
Title: Impact of the Oral Microbiota on Relapse in HNSCC Patients
Acronym: MICR-ORL
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Sainte Catherine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MICR-ORL
Record Dates: First submitted 2025-01-20; First posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- buccal swabs (Experimental): buccal swabs for microbiota analysis before and after treatment
  Interventions: Other: buccal swabs

INTERVENTIONS:
Other: buccal swabs — buccal swabs for microbiota analysis before and after radiotherapy

SUMMARY:
to characterise the impact of microbiota in radiotherapy efficacy

ELIGIBILITY:
Inclusion Criteria:

* head and neck cancer

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2027-01-20 (Estimated)

PRIMARY OUTCOMES:
Microbiota | 2 years
  Analysis of buccal microbiota by 16SrRNA gene sequencing

CONTACTS AND LOCATIONS:
Locations (1):
- ICAP, Avignon, France

IPD SHARING:
Plan to Share IPD: No